CLINICAL TRIAL: NCT07283042
Title: Evaluation of Clinical Outcomes and Acceptability of an Anatomical Classification for Placenta Accreta
Brief Title: Evaluation of Clinical Outcomes and Acceptability of an Anatomical Classification for Placenta Accreta Spectrum
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Yalda Afshar, MD, PhD, Professor of Obstetrics and Gynecology, University of California, Los Angeles
Other Study IDs: 24-6300
Record Dates: First submitted 2025-11-19; First posted 2025-12-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal Blood, Cord Blood, Cord Biopsy, and Placental Biopsy will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PAS: Patients with placental accreta undergoing planned surgical intervention for PAS
  Interventions: Procedure: Total Hysterectomy; Procedure: Modified subtotal hysterectomy; Procedure: One-Step Conservative Surgery

INTERVENTIONS:
Procedure: Total Hysterectomy — Removal of entire uterus
Procedure: Modified subtotal hysterectomy — When partial tissue integrity is preserved
Procedure: One-Step Conservative Surgery — Considered when significant healthy myometrium is preserved

SUMMARY:
This study evaluates the clinical implementation of intra-operative topographic classification system for PAS. In addition to a standard of care risk stratification prenatal ultrasound for patients with a risk of PAS, this study adds an additional intraoperative surgical staging protocol to validate the classification system, improve surgical approach, and significantly clinical outcomes of pregnant people with an a prior risk of PAS. The study will involve pregnant patients with PAS risk factor, include data collection spanning prenatal assessment, intraoperative classification, surgical technique implementation and postoperative analysis. The anticipated study duration is approximately 36-48 months.

DETAILED DESCRIPTION:
This study is a prospective cohort study designed to assess the validity, feasibility, and clinical utility of a topographic classification system for placenta accreta spectrum (PAS), with a primary focus on its application in the actual execution of surgery. This study is investigating a clinical decision flowchart used for intraoperative staging and classification of placenta accreta spectrum (PAS) or similar uterine surgical scenarios. It integrates topographic classification, surgical decision-making, and treatment strategy selection.

The classification system will directly guide and be integrated into real-time surgical planning and management-from cesarean hysterectomy to one-step conservative surgery-based on prenatal ultrasound staging and intraoperative findings.

* Standardizing prenatal ultrasound staging for PAS.
* Implementing a structured protocol for intraoperative classification and surgical execution according to ultrasound.
* Collecting and correlating surgical and pathological findings, including intraoperative photos, videos, and gross and histological analysis.
* Utilizing an objective method to quantify intraoperative blood loss.
* Comparing preoperative ultrasound findings with intraoperative and postoperative data to validate the classification system.
* Managing participant dropouts and protocol deviations to ensure data integrity and minimize bias.
* Applying appropriate statistical adjustments for multiple group comparisons to reduce the risk of type I error. Methods such as Bonferroni correction or false discovery rate adjustments will be utilized where applicable.
* Incorporating serial blood draws for plasma and whole blood analysis to identify potential biomarkers associated with PAS severity, surgical complexity, and clinical outcomes. This will be optional and stored in the biorepository.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant people suspected of having PAS based on ultrasound findings or clinical risk factors
* Patients undergoing planned surgical intervention for PAS, including a planned cesarean
* Individuals who provide informed consent to participate in the study
* Patients with at least one prenatal assessment before surgery
* Expected age range: 18-55
* Patient has agreed to conservative management approach as part of standard of care if feasible intraoperatively

Exclusion Criteria:

* Patients who decline participation or withdraw consent
* Those with contraindications to the planned surgical procedure

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be comprised of pregnant people suspected of having PAS. PAS is a major obstetric complication associated with significant maternal morbidity and mortality that is increasing in prevalence due to the rising rate of cesarean births, which are the biggest clinical risk factor
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound assessment | 0-30 days prior to planned surgery
  Prenatal ultrasound assessment using the "Ultrasound Staging" protocol (6 views), with classification into one of the topographic categories
Surgical Procedure and Classification | At time of surgery
  Intraoperative classification of the placental lesion using the topographic classification system
Quantification of Blood Loss | Documented throughout surgery and at the completion of the procedure
  Objective quantification of blood loss using suction devices, surgical sponges, and vaginal bleeding
Gross Pathological Analysis of Resected Tissues | Within 2 hours post surgery
  Post-surgery gross pathological analysis of resected tissues to correlate with ultrasound and surgical findings
Adverse Events | Up to 12 months post surgery
  Presence of any of the following during follow up will be measured in a binary fashion (Yes/No): re-admissions, re-operations, infection/sepsis, wound seroma.

CONTACTS AND LOCATIONS:
Overall Officials: Yalda Afshar, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No